CLINICAL TRIAL: NCT01314287
Title: Observational Study of the Effect of Coughing on Emergence From Anaesthesia on Oxygenation in the Postanaesthetic Care Unit
Brief Title: Effect of Coughing on Oxygenation in the Post Anaesthetic Care Unit
Status: Completed | Type: Observational
Sponsor: NHS Research and Development (Other Government)
Collaborators: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Andrew Lumb, Consultant Anaesthetist, NHS Research and Development
Other Study IDs: AN10/9556; 10/H1307/127 (Other: Leeds West REC)
Record Dates: First submitted 2011-03-11; First posted 2011-03-14 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-04

CONDITIONS: Adverse Effect of Unspecified General Anesthetics
Keywords: Anaesthesia; pulmonary complications; Atelectasis
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
General anaesthesia causes small areas of lung to collapse (referred to as atelectasis) and many strategies are used to prevent or reverse this, but these strategies only temporarily improve lung function and do not persist into the post anaesthesia care unit (PACU) where atelectasis may still be present. One possible explanation for this is that coughing occurring at the end of the anaesthesic may cause atelectasis to occur. Over 70% of patients cough when their breathing tube is removed as they emerge from the anaesthetic, and our hypothesis is that the presence of the breathing tube prevents a normal cough from occurring and may worsen atelectasis. This study will use alveolar-arterial oxygen difference (AaDO2)as a measure of how well the lungs are oxygenating the blood. This will be measured 30 minutes before the end of the anaesthetic as a control measure of the patient's lung function, and again 60 minutes after the patient has woken up, and the change compared with the amount of coughing observed as the patient emerges from the anaesthetic.

DETAILED DESCRIPTION:
This is an observational study which hopes to answer the question of whether the amount of coughing that occurs when a patient emerges from anaesthesia has a negative impact on the ability of the lung to transfer oxygen to the blood in the post anaesthetic care unit (PACU). The patients' involvement starts 45 minutes before the anticipated end of surgery when a standard lung recruitment manoevre will be performed. Fifteen minutes later a 2ml blood sample is taken from the arterial catheter which was placed at the beginning of surgery. From this, together with routinely monitored clinical data, the alveolar/arterial oxygen difference (AaDO2) is calculated. The AaDO2 is used as a measure of the degree of impairment of the lung's ability to fully oxygenate the blood. Next, as the patient wakes up from the anaesthesia, an observer (who is not involved in the clinical care of the patient) will record the amount of coughing that occurs. Assessment of coughing will involve recording:

* time spent coughing
* the number of coughs before and after removing the breathing tube Postoperative care will be routine with oxygen given as required. 1 hour after removal of the tracheal tube a second arterial blood sample is taken from the arterial catheter whilst the patient is breathing 40% oxygen and once again the AaDO2 is calculated. Following the second blood sample the subject's involvement with the study ends.

During the operation no stipulations are made regarding the anaesthetic technique to be used, which is left entirely at the discretion of the anaesthetist with clinical responsibility for the patient. In the last 30 minutes of the operation, the patient's artificial ventilation will be with an oxygen concentration of 40% and a set 'positive end expiratory pressure'(PEEP). Other than that, anaesthetists will be free to wake the patient up by their own preferred method. Also, if at any time the responsible anaesthetist feels the adjustment of the ventilation is required in order to act in the patient's best interest, the patient will be removed from the trial.

Data to be recorded will include sex, age, ASA grade (a measurement of the patients' fitness for an anaesthetic), height and weight, whether or not the patient is a smoker and whether the patient has any lung disease. At the end of surgery, the operation performed and its duration will be recorded. These data are required to characterise the population of patients studied and allow comparison with other research.

No medication or perioperative treatment need be withheld or modified as a consequence of the patient being enrolled in the study. There is no requirement for starting any addition medication as a consequence of the study. Patients may withdraw at any time by withdrawal of consent, in which case all subject data will be destroyed and only the fact that consent was withdrawn will be documented. The anaesthetist with clinical responsibility for the patient may withdraw the patient from the study at any time, in which case the reason for withdrawal will be documented on the data collection form and any data collected will be kept until study completion.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be selected who require, as part of their normal clinical anaesthetic care, a breathing tube in their lungs and a small plastic tube (catheter) placed in an artery for monitoring and blood sampling

Exclusion Criteria:

* Refusal or inability to provide written, informed consent
* Respiratory disease which is severe enough to prevent the safe use of the oxygen levels required for this study
* A expectation that the patient will require their breathing to be supported artificially after the operation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study subjects will be adult patients undergoing routine operations which are expected to last longer than 45 minutes.
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2011-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change in oxygenation before and after emergence from general anaesthesia | 2 hours
  Change between intraoperative and postoperative AaDO2 for each patient in relation to the amount of coughing observed on emergence from anaesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew B Lumb, MB BS FRCA, Principal Investigator — Leeds Teaching Hospitals NHS Trust
Locations (1):
- St James's University Hospital, Leeds, West Yorkshire, United Kingdom